CLINICAL TRIAL: NCT05914090
Title: The Application of Enhanced Recovery After Surgery (ERAS) for Cardiovascular Surgery in Adult: a Stepped Wedge Cluster Randomized Trial
Brief Title: The Application of Enhanced Recovery After Surgery (ERAS) for Cardiovascular Surgery in Adult
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yan Fuxia (Other)
Responsible Party: Sponsor-Investigator, Yan Fuxia, principal investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023--1968
Record Dates: First submitted 2023-05-15; First posted 2023-06-22 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Surgery; Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Procedure: ERAS
- Control group (No Intervention)

INTERVENTIONS:
Procedure: ERAS — Among adults, patients undergoing elective extracorporeal circulation for cardiac surgery are included in the ERAS strategy intervention plan, which mainly includes preoperative education, preoperative oral intake of multidimensional carbohydrate beverages, multimodal analgesia, blood protection strategies, correction of perioperative hypoalbuminemia, early removal of tracheal intubation, maintenance of blood sugar at reasonable levels, and targeted liquid therapy.
  Arms: Intervention group

SUMMARY:
Among adults, patients undergoing elective extracorporeal circulation for cardiac surgery are included in the ERAS strategy intervention plan, which mainly includes preoperative education, preoperative oral intake of multidimensional carbohydrate beverages, multimodal analgesia, blood protection strategies, correction of perioperative hypoalbuminemia, early removal of tracheal intubation, maintenance of blood sugar at reasonable levels, and targeted liquid therapy. The traditional plan group follows the current clinical diagnosis and treatment routine. By comparing the differences in the incidence of major postoperative outcomes (MACCE events, major pulmonary complications, and acute kidney injury) between the intervention group and the non intervention group, as well as comparing other adverse events (including but not limited to pneumonia, massive bleeding, postoperative arrhythmia, incision infection, postoperative nausea, vomiting, and delirium), all cause secondary intubation, and all cause secondary surgery between the two groups, and recording hospitalization time, ICU stay time The removal time of tracheal intubation and drainage tube, as well as the pain score during hospitalization and the total amount of opioid drug use (converted to equivalent dose morphine), hospitalization cost, postoperative recovery quality QoR15 scale score, and patient satisfaction score, were recorded to explore whether the ERAS regimen can reduce the incidence of major postoperative adverse events, improve patient prognosis, and accelerate postoperative recovery compared to traditional regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years
* Patients awaiting elective cardiac surgery with cardiopulmonary bypass (CPB)

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) class is above class V
* Patients with cardiac assist device or mechanical ventilation
* The ejection fraction of patients is less than 30%
* Patients with morbid obesity
* Patients with severe obstructive sleep apnea-hypopnea syndrome (OSAHS)
* Patients with severe pulmonary disease, including severe chronic obstructive pulmonary disease (COPD) or respiratory failure
* Patients with severe liver or renal dysfunction, including severe acute or chronic renal dysfunction need renal replacement therapy, and acute or chronic liver failure need artificial liver therapy
* Patients with long-term opioid or sedative utilization
* Patients with a history of alcohol or cigarette abuse
* Patients with long-term hormone therapy
* An international normalized ratio > 2.0
* Patients with severe malnutrition
* Mental or legal disability
* Current enrollment in another clinical trial
* Patients' refusal or low adherence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2023-10-11 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcomes | during hospitalization, an average of 1 week, assessed up to 30 days
  The composite outcomes include the major adverse cardiac and cerebrovascular events (MACCE), major postoperative pulmonary complication (PPCs), and acute kidney injury (AKI).

SECONDARY OUTCOMES:
the quality of recovery score (QoR)-15 after surgery | At 24 hour after surgery
length of hospital stay | From the date of admission until the date of discharging, assessed up to 30 days
  From the date of admission until the date of discharging
the duration of intensive care unit (ICU) stay | Time from ICU admission to ICU discharge, assessed up to 30 days
  Time from ICU admission to ICU discharge
time to extubation | The time from the end of operation to the removal of tracheal intubation, assessed up to 30 days
  The time from the end of operation to the removal of tracheal intubation
time to drainage removal | The time from the end of operation to the removal of drainage tube, assessed up to 30 days
  The time from the end of operation to the removal of drainage tube
the rate of other complications | during hospitalization, an average of 1 week, assessed up to 30 days
  The rate of other complications include delium, pneumonia, pneumothorax, hematorrhea and so on
the rate of reintubation for any cause | during hospitalization, an average of 1 week, assessed up to 30 days
  The rate of reintubation for any cause
cumulative opioid dosage | during hospitalization, an average of 1 week, assessed up to 30 days
  Total perioperative consumption of opioid analgesics
overall medical costs | during hospitalization, an average of 1 week, assessed up to 30 days
  Total cost of patients during hospitalization
satisfaction score | the day before discharge, assessed up to 30 days
  A satisfaction rating using a 0-10 number scale (0=unsatisfactory, 10=satisfactory)
the outcomes of long-term prognosis by telephone follow-up | within 30 days, 3 months, and 1 year
  the outcomes of prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, China, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No